CLINICAL TRIAL: NCT05923372
Title: Evaluation of the Disability-Adjusted Life Year (DALY) on a Cohort of Patients With Indolent Systemic Mastocytosis (ISM)
Brief Title: Evaluation of the DALY on a Cohort of Patients With Indolent Systemic Mastocytosis
Acronym: DALY-MAST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/23/0011; 2023-A00178-37 (Other: N°ID-RCB)
Record Dates: First submitted 2023-06-19; First posted 2023-06-28 (Actual); Last update posted 2023-07-12 (Actual); Status verified 2023-07

CONDITIONS: Mastocytosis, Indolent Systemic
Keywords: DALY; Mastocytosis; Quality of life
MeSH Terms: conditions — Mastocytosis, Systemic; Mastocytosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with indolent systemic mastocytosis (IMS): Patients with IMS, included in the CEREMAST registry and who have given their consent to participate

SUMMARY:
Mastocytosis is a group of pathologies characterized by the accumulation and/or clonal proliferation of abnormal mast cells in various organs. The impact of mastocytosis on health, quality of life, the psychoaffective sphere and on professional life constitutes the burden of this disease. The DALY is the disability-adjusted life expectancy, which takes into account the life expectancy and the number of years "lost" due to illness, disability or early death. Due to the major impact of the disease this study evaluates the DALY in indolent mastocytosis patients

DETAILED DESCRIPTION:
Mastocytosis is a group of pathologies characterized by the accumulation and/or clonal proliferation of abnormal mast cells in various organs. Mastocytosis is a rare disease with an estimated prevalence of between 1/20,000 and 1/40,000. The impact of mastocytosis on health, quality of life, the psychoaffective sphere and on professional life constitutes the burden of this disease. This is probably important but very little studied so far. The DALY is the disability-adjusted life expectancy. It is calculated by subtracting from life expectancy the number of years "lost" due to illness, disability or early death.

Ignorance of the disease and diagnostic error cause significant distress in patients. In our clinical experience, the impact of the disease on the personal, social, and professional life of our patients is major. It therefore seems important to better specify the impact on the quality of life and the costs of this pathology. The main objective of this study is to evaluate the DALY in indolent mastocytosis patients from the CEREMAST reference center of the Toulouse University Hospital.

ELIGIBILITY:
Inclusion Criteria:

* Having expressed their non opposition to participate in this study
* Diagnosed with indolent mastocytosis and cared for in the CEREMAST reference center in Toulouse

Exclusion Criteria:

* Patient with a form of mastocytosis other than MSI
* Patient under legal protection, guardianship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with MSI, included in the CEREMAST register and who have given their consent to participate
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
DALY | Day 1
  DALY (Disability Adjusted Life Year): Its calculation consists of subtracting from life expectancy the number of years "lost" due to illness, disability or early death.

SECONDARY OUTCOMES:
Quality of life based on the MC QOL scale | Day 1
  The quality of life of the included patients will be described with the The Mastocytosis Quality of Life Questionnaire (MC-QoL) which has scores from 0 to 100, where higher scores indicate higher health-related quality-of-life impairment
Frequency of symptoms | Day 1
  The frequency of various symptoms of mast cell activation will also be described.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina BULAI LIVIDEANU, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- Centre de Référence des Mastocytoses, Service de Dermatologie, Hôpital Larrey, CHU Toulouse, Toulouse, Haute-Garonne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siebenhaar F, Fortsch A, Krause K, Weller K, Metz M, Magerl M, Martus P, Church MK, Maurer M. Rupatadine improves quality of life in mastocytosis: a randomized, double-blind, placebo-controlled trial. Allergy. 2013 Jul;68(7):949-52. doi: 10.1111/all.12159. Epub 2013 Jun 4. PMID 23734572
- [Background] Siebenhaar F, von Tschirnhaus E, Hartmann K, Rabenhorst A, Staubach P, Peveling-Oberhag A, Wagner N, Martus P, Carter MC, Metcalfe DD, Church MK, Maurer M, Weller K. Development and validation of the mastocytosis quality of life questionnaire: MC-QoL. Allergy. 2016 Jun;71(6):869-77. doi: 10.1111/all.12842. Epub 2016 Feb 15. PMID 26797792
- [Background] van Anrooij B, Kluin-Nelemans JC, Safy M, Flokstra-de Blok BM, Oude Elberink JN. Patient-reported disease-specific quality-of-life and symptom severity in systemic mastocytosis. Allergy. 2016 Nov;71(11):1585-1593. doi: 10.1111/all.12920. Epub 2016 Jun 23. PMID 27089859
- [Background] Jennings SV, Slee VM, Zack RM, Verstovsek S, George TI, Shi H, Lee P, Castells MC. Patient Perceptions in Mast Cell Disorders. Immunol Allergy Clin North Am. 2018 Aug;38(3):505-525. doi: 10.1016/j.iac.2018.04.006. PMID 30007467
- [Background] Jennings S, Russell N, Jennings B, Slee V, Sterling L, Castells M, Valent P, Akin C. The Mastocytosis Society survey on mast cell disorders: patient experiences and perceptions. J Allergy Clin Immunol Pract. 2014 Jan-Feb;2(1):70-6. doi: 10.1016/j.jaip.2013.09.004. Epub 2013 Dec 3. PMID 24565772
- [Background] Nowak A, Gibbs BF, Amon U. Pre-inpatient evaluation on quality and impact of care in systemic mastocytosis and the influence of hospital stay periods from the perspective of patients: a pilot study. J Dtsch Dermatol Ges. 2011 Jul;9(7):525-32. doi: 10.1111/j.1610-0387.2011.07638.x. Epub 2011 Mar 24. English, German. PMID 21992665
- [Background] Sanchez-Munoz L, Morgado JM, Alvarez-Twose I, Matito A, Garcia-Montero AC, Teodosio C, Jara-Acevedo M, Mayado A, Mollejo M, Caldas C, Gonzalez de Olano D, Escribano L, Orfao A. Diagnosis and classification of mastocytosis in non-specialized versus reference centres: a Spanish Network on Mastocytosis (REMA) study on 122 patients. Br J Haematol. 2016 Jan;172(1):56-63. doi: 10.1111/bjh.13789. Epub 2015 Oct 12. PMID 26456532
- [Background] Jackson CW, Pratt CM, Rupprecht CP, Pattanaik D, Krishnaswamy G. Mastocytosis and Mast Cell Activation Disorders: Clearing the Air. Int J Mol Sci. 2021 Oct 19;22(20):11270. doi: 10.3390/ijms222011270. PMID 34681933
- [Background] Valent P, Horny HP, Escribano L, Longley BJ, Li CY, Schwartz LB, Marone G, Nunez R, Akin C, Sotlar K, Sperr WR, Wolff K, Brunning RD, Parwaresch RM, Austen KF, Lennert K, Metcalfe DD, Vardiman JW, Bennett JM. Diagnostic criteria and classification of mastocytosis: a consensus proposal. Leuk Res. 2001 Jul;25(7):603-25. doi: 10.1016/s0145-2126(01)00038-8. PMID 11377686
- [Background] Afrin LB. Mast cell activation disease and the modern epidemic of chronic inflammatory disease. Transl Res. 2016 Aug;174:33-59. doi: 10.1016/j.trsl.2016.01.003. Epub 2016 Jan 18. PMID 26850903
- [Background] Hermouet S, Bigot-Corbel E, Gardie B. Pathogenesis of Myeloproliferative Neoplasms: Role and Mechanisms of Chronic Inflammation. Mediators Inflamm. 2015;2015:145293. doi: 10.1155/2015/145293. Epub 2015 Oct 11. PMID 26538820